CLINICAL TRIAL: NCT03460587
Title: Long-term Telerehabilitation for Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Steven C. Cramer, MD, Professor of Neurology, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17IRG3346039
Record Dates: First submitted 2018-02-28; First posted 2018-03-09 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-06

CONDITIONS: Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Home-based Telerehabilitation (Experimental): Home-based Telerehabilitation
  Interventions: Device: Telerehabilitation

INTERVENTIONS:
Device: Telerehabilitation — The Telerehabilitation system will deliver rehabilitation treatment sessions via an in-home internet-connected computer. A major component of the system is the use of games to promote therapeutically relevant movements. The subject will perform daily assigned home-based telerehabilitation games and exercises and 5 minutes of stroke education, all guided by the telerehabilitation system.During some of the sessions, therapists will initiate a videoconference with the subject's telerehabilitation system to discuss progress, issues, and revise treatment plans as needed.

SUMMARY:
The aim of the current protocol is to study 40 patients, each for 12 weeks, to address hypotheses related to the ability of a telerehabilitation system to (a) improve motor status and disability, (b) collect various forms of patient data from the home, (c) improve risk factor knowledge and control, and (d) assess patient compliance with home-based telerehabilitation.

Patients who have returned to their home after stroke will be provided with a telehealth system and be asked to use it 6 days/week for 12 weeks, during which time subjects will use this system for daily rehabilitation therapy, assessments, and education--all on one platform.

DETAILED DESCRIPTION:
Stroke is perennially one of the leading causes of human disability. Stroke is truly a chronic disease, with survivors living for years or decades after the event. Increasing evidence describes years of steady decline in several health measures for stroke survivors. Many factors contribute to this, including further strokes, uncontrolled risk factors, development of late complications of stroke, and limited access to rehabilitation therapy.

New approaches are needed that address the many needs of stroke survivors, efficiently and in aggregate. Emerging telehealth technologies have high potential to address this major unmet need, but substantial innovation will be needed. The long-term goal is to establish a telehealth platform to treat chronic stroke.

A telehealth system will be delivered to enrollee's home. Patients will be asked to interact with their system daily (at least 6 days/wk) for 12 weeks. For 3 times per week, during the first 2 weeks, and then 1 time per week thereafter, a study therapist or research assistant in the lab will use the telehealth system to have a videoconference with the subject, to answer questions, provide feedback, review progress, and make any changes needed in the therapy plan. Study personnel will monitor usage statistics and performance measures for all systems.

A key strategy is to measure in parallel, patient behaviors in three categories of health issues central to chronic stroke: (1) medical management issues including risk factor knowledge and control, (2) disability issues including motor function, and (3) psychological issues including depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of randomization
2. Stroke that is radiologically verified, due to ischemia or to intracerebral hemorrhage or subarachnoid hemorrhage, and with any time of stroke onset prior to randomization
3. Arm motor Fugl Meyer score of 28-66; if Arm motor Fugl Meyer score> 59, must also have Box & Blocks on affected side >25% lower
4. Box & Block Test score with affected arm is at least 3 blocks in 60 seconds at the first visit
5. Informed consent signed by the subject
6. Behavioral contract signed by the subject

Exclusion Criteria:

1. A major, active, coexistent neurological or psychiatric disease, including alcoholism or dementia
2. A diagnosis (apart from the index stroke) that substantially affects paretic arm function
3. A major medical disorder that substantially reduces the likelihood that a subject will be able to comply with all study procedures
4. Severe depression, defined as Geriatric Depression Scale Score >11
5. Significant cognitive impairment, defined as Montreal Cognitive Assessment score < 22; note that this exclusion criteria can be waived at the discretion of the study PI, e.g., for aphasia
6. Deficits in communication that interfere with reasonable study participation
7. Lacking visual acuity, with or without corrective lens, of 20/40 or better in at least one eye
8. Life expectancy < 6 months
9. Receipt of Botox to arms, legs, or trunk in the preceding 6 months, or expectation that Botox will be administered to the arm, leg, or trunk prior to completion of participation in this study
10. Unable to successfully perform all 3 of the rehabilitation exercise test examples
11. Unable or unwilling to perform study procedures/therapy, or expectation of non-compliance with study procedures/therapy, or expectation that subject will be unable to participate in study visits
12. Concurrent enrollment in another investigational study
13. Non-English speaking, such that subject does not speak sufficient English to comply with study procedures
14. Expectation that subject will not have a single domicile address during the 12 weeks of therapy, within 75 miles of the central study site
15. Note that the presence of wireless home internet connectivity is not an exclusion criterion, but preference may be given to enrollees who do have wireless home internet connectivity because this will enable testing of study hypotheses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cramer, MD, Principal Investigator — UC Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dodakian L, McKenzie AL, Le V, See J, Pearson-Fuhrhop K, Burke Quinlan E, Zhou RJ, Augsberger R, Tran XA, Friedman N, Reinkensmeyer DJ, Cramer SC. A Home-Based Telerehabilitation Program for Patients With Stroke. Neurorehabil Neural Repair. 2017 Oct-Nov;31(10-11):923-933. doi: 10.1177/1545968317733818. Epub 2017 Oct 26. PMID 29072556
- [Background] Cramer SC, Sur M, Dobkin BH, O'Brien C, Sanger TD, Trojanowski JQ, Rumsey JM, Hicks R, Cameron J, Chen D, Chen WG, Cohen LG, deCharms C, Duffy CJ, Eden GF, Fetz EE, Filart R, Freund M, Grant SJ, Haber S, Kalivas PW, Kolb B, Kramer AF, Lynch M, Mayberg HS, McQuillen PS, Nitkin R, Pascual-Leone A, Reuter-Lorenz P, Schiff N, Sharma A, Shekim L, Stryker M, Sullivan EV, Vinogradov S. Harnessing neuroplasticity for clinical applications. Brain. 2011 Jun;134(Pt 6):1591-609. doi: 10.1093/brain/awr039. Epub 2011 Apr 10. PMID 21482550
- [Background] Kwakkel G, Wagenaar RC, Twisk JW, Lankhorst GJ, Koetsier JC. Intensity of leg and arm training after primary middle-cerebral-artery stroke: a randomised trial. Lancet. 1999 Jul 17;354(9174):191-6. doi: 10.1016/S0140-6736(98)09477-X. PMID 10421300
- [Derived] Cramer SC, Dodakian L, Le V, McKenzie A, See J, Augsburger R, Zhou RJ, Raefsky SM, Nguyen T, Vanderschelden B, Wong G, Bandak D, Nazarzai L, Dhand A, Scacchi W, Heckhausen J. A Feasibility Study of Expanded Home-Based Telerehabilitation After Stroke. Front Neurol. 2021 Feb 3;11:611453. doi: 10.3389/fneur.2020.611453. eCollection 2020. PMID 33613417

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Home-based Telerehabilitation
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients who signed informed consent.
Arm/Group | Home-based Telerehabilitation
Number analyzed (Participants) | 13
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [52 to 65.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Time post-stroke [Median (Inter-Quartile Range); unit: days] | 129 [52 to 486]
Arm motor Fugl-Meyer score [Median (Inter-Quartile Range); unit: units on a scale] | 46 [42 to 57]
Leg motor Fugl-Meyer score [Median (Inter-Quartile Range); unit: units on a scale] | 28 [23.5 to 29]

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Arm Motor Scale
Description: measure of arm impairment, scores range from 0 to 66 with higher numbers reflecting less arm impairment
Time Frame: 90 days
Population: All patients who signed informed consent.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Home-based Telerehabilitation
Number analyzed (Participants) | 13
units on a scale | 59 [52.5 to 61.5]

2. Secondary Outcome: Fugl-Meyer Leg Motor Scale
Description: measure of leg impairment, scores range from 0 to 34 with higher numbers reflecting less leg impairment
Time Frame: 90 days
Population: All patients who signed informed consent
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Home-based Telerehabilitation
Number analyzed (Participants) | 13
units on a scale | 28 [27 to 30.5]

ADVERSE EVENTS:
Time Frame: From enrollment to 90 days later
Description: All adverse events and serious adverse events were recorded.
Arm/Group | Home-based Telerehabilitation
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT03460587/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT03460587/SAP_001.pdf